CLINICAL TRIAL: NCT06141265
Title: Chemotherapy Combined With Bevacizumab Followed by Niraparib Monotherapy in Newly Diagnostic Advanced Ovarian Cancer With HRD Positive : A Perspective, Multicenter, Single-arm Phase II Trial
Brief Title: Niraparib Maintenance in HRD-Positive Advanced Ovarian Cancer Following Front-Line Chemotherapy + Bevacizumab
Acronym: BRAND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hong Zheng, M.D., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YJZ62
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib (Experimental): The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count

SUMMARY:
This study is a multicenter, open-label, single-arm phase II clinical trial investigating the efficacy and safety of niraparib monotherapy maintenance in HRD-positive newly diagnosed advanced epithelial ovarian cancer (EOC), including primary peritoneal and/or fallopian tube tumors, following response to front-line chemotherapy in combination with bevacizumab. A total of 116 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. The written informed consent form shall be signed before proceeding with any study-related procedure.
2. Participants shall be a female, aged 18 years or older.
3. Histologically confirmed primary high-grade epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma。
4. FIGO staging is Stage III or IV.
5. Patients who have undergone primary tumor reductive surgery or intermittent tumor reductive surgery (patients who have used neoadjuvant therapy), regardless of postoperative residual lesion status
6. Participants must have received, prior to enrollment, a minimum of 2 cycles of bevacizumab in combination with platinum-based chemotherapy.
7. Participants must have completed front-line, platinum-based chemotherapy with CR, PR, or NED assessed by RECIST v1.1.
8. Participant must have either CA-125 in the normal range or CA-125 decrease by more than 90% during front-line therapy that is stable for at least 7 days (ie, no increase > 15% from nadir).
9. Participants must have first study treatment dose within 12 weeks of the first day of the last cycle of chemotherapy.
10. Genetic testing of tumor tissue indicates HRD positive or germline/somatic BRCA mutation prior to enrollment.
11. Participant must have an Eastern Cooperative Oncology Group (ECOG) score ≤2.
12. Organ function is in good condition, including: Hemoglobin ≥100 g/L; White blood cell count ≥3×10^9/L; Neutrophil count ≥1.5×10^9/L; Platelet count ≥100×10^9/L; Total bilirubin is not more than 1.5 times the normal upper limit; ALK, AST and ALT are not more than 2.5 times their normal upper limit, and with existence of hepatic metastasis, these values must not be more than 5 times their normal upper limit; Serum creatinine is not more than 1.5 times the normal upper limit.

Exclusion Criteria:

1. Histopathological types other than high-grade ovarian/tubal/peritoneal cancer or metastatic ovarian cancer.
2. Receipt of other targeted drugs as maintenance therapy, excluding PARP inhibitors.
3. Concurrent severe respiratory or hematologic disorders, poorly controlled diabetes, uncontrolled hypertension of Grade 2 or higher, NYHA Class III or higher congestive heart failure, unstable angina, recent myocardial infarction within the past 6 months, or other circulatory system diseases.
4. Any other significant complications or functional impairments in organ systems, as determined by the investigator, that may affect the safety of the participant or interfere with the evaluation of the investigational drug.
5. Expected survival less than 3 months.
6. Other than ovarian cancer, the participant has been diagnosed a second primary tumor within the past 2 years and currently undergoing treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) Rate at 24 months (PFS24) | At 24 months
  PFS rate at 24 months is defined as the percentage of participants who have not progressed or died within 24 months after niraparib treatment initiation. Progression was assessed by response evaluation criteria in solid tumors (RECIST) version (v) 1.1 criteria per Investigator assessment. Survival rate is the percentage of participants without progression assessed by RECIST v1.1 or death by the landmark timepoint. Confidence intervals was constructed using exact method.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) Rate at 12 months (PFS12) | At 12 months
  PFS rate at 12 months after niraparib treatment initiation according to investigator assessment
Time to First Subsequent Therapy (TFST) | up to 36 months
  Time from the date of initiation of maintenance therapy with niraparib to the date of the first subsequent anticancer therapy or death, whichever occurred first.
Time to Second Subsequent Therapy (TSST) | up to 48 months
  Time from the date of initiation of maintenance therapy with niraparib to the date of the second subsequent anticancer therapy or death, whichever occurred first.
Median Progression Free Survival（mPFS） | up to 36 months
  Time from the date of initiation of maintenance therapy with niraparib to the date of disease progression in our study

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No